CLINICAL TRIAL: NCT00010283
Title: Oral Beclomethasone Dipropionate Capsules for Treatment of Intestinal Graft-Versus-Host Disease: Compassionate Use in Patients With Contraindictions to High-Dose Immunosuppressive Therapy
Brief Title: Beclomethasone in Treating Patients With Graft-Versus-Host Disease of the Esophagus, Stomach, Small Intestine, or Colon
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: 1500.00; FHCRC-1500.00; RPCI-DS-99-27; NCI-H01-0067; CDR0000068475 (Registry Identifier: PDQ)
Record Dates: First submitted 2001-02-02; First posted 2004-04-13 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-03

CONDITIONS: Breast Cancer; Chronic Myeloproliferative Disorders; Gestational Trophoblastic Tumor; Graft Versus Host Disease; Kidney Cancer; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Neuroblastoma; Ovarian Cancer; Testicular Germ Cell Tumor
Keywords: stage III breast cancer; stage IV breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; Burkitt lymphoma; extramedullary plasmacytoma; refractory multiple myeloma; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; disseminated neuroblastoma; recurrent neuroblastoma; recurrent Wilms tumor and other childhood kidney tumors; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; recurrent childhood lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; stage III malignant testicular germ cell tumor; childhood diffuse large cell lymphoma; recurrent malignant testicular germ cell tumor; childhood immunoblastic large cell lymphoma; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; chronic idiopathic myelofibrosis; essential thrombocythemia; testicular embryonal carcinoma; testicular choriocarcinoma; testicular teratoma; testicular yolk sac tumor; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and teratoma with seminoma; testicular embryonal carcinoma and yolk sac tumor; testicular embryonal carcinoma and yolk sac tumor with seminoma; testicular embryonal carcinoma and seminoma; testicular yolk sac tumor and teratoma; testicular yolk sac tumor and teratoma with seminoma; testicular choriocarcinoma and yolk sac tumor; testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and teratoma; testicular choriocarcinoma and seminoma; refractory hairy cell leukemia; recurrent/refractory childhood Hodgkin lymphoma; recurrent ovarian germ cell tumor; chronic myelomonocytic leukemia; ovarian yolk sac tumor; ovarian embryonal carcinoma; ovarian polyembryoma; ovarian choriocarcinoma; ovarian immature teratoma; ovarian mature teratoma; ovarian monodermal and highly specialized teratoma; ovarian mixed germ cell tumor; acute undifferentiated leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; poor prognosis metastatic gestational trophoblastic tumor; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; graft versus host disease; prolymphocytic leukemia; primary systemic amyloidosis; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; anaplastic large cell lymphoma; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Breast Neoplasms; Myeloproliferative Disorders; Gestational Trophoblastic Disease; Graft vs Host Disease; Kidney Neoplasms; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Neuroblastoma; Ovarian Neoplasms; Testicular Germ Cell Tumor; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Burkitt Lymphoma; Carcinoma, Ovarian Epithelial; Wilms Tumor; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Testicular Neoplasms; Lymphoma, Large B-Cell, Diffuse; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Primary Myelofibrosis; Thrombocythemia, Essential; Teratoma, Testicular; Endodermal Sinus Tumor; Teratoma; Seminoma; Carcinoma, Embryonal; Leukemia, Hairy Cell; Recurrence; Leukemia, Myelomonocytic, Chronic; Leukemia, Biphenotypic, Acute; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Immunoglobulin Light-chain Amyloidosis; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone | interventions — Beclomethasone

INTERVENTIONS:
Drug: beclomethasone dipropionate

SUMMARY:
RATIONALE: Beclomethasone may be an effective treatment for graft-versus-host disease.

PURPOSE: Phase I/II trial to study the effectiveness of beclomethasone in treating patients who have graft-versus-host disease of the esophagus, stomach, small intestine, or colon.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the frequency of treatment success in patients with intestinal graft-versus-host disease with contraindications to high-dose immunosuppressive therapy treated with beclomethasone. II. Determine the frequency of adverse events related to the use of this drug in these patients. III. Assess the natural history and outcome of the medical problem for which high-dose immunosuppressive therapy was a contraindication.

OUTLINE: Patients receive oral beclomethasone 4 times daily for 28 days. Treatment may repeat for an additional 28 days as needed. Patients are interviewed weekly to assess treatment success and adverse events. Patients are followed at 1 and 2 weeks.

PROJECTED ACCRUAL: A total of 40-100 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven intestinal (esophagus, stomach, small intestine, or colon) graft-versus-host disease (GVHD) exhibiting symptoms such as nausea, vomiting, anorexia, diarrhea, or abdominal pain in the absence of another explanation for these symptoms Specific contraindications to high-dose immunosuppressive therapy, such as: Recurrent malignant disorder for which an allogeneic antitumor effect is desired Aspergillus or other fungal infection Severe myopathy, hyperglycemia, bone problems, or neuropsychiatric symptoms related to corticosteroid use Thrombotic thrombocytopenic purpura or hemolytic uremic syndrome related to immunosuppressive therapy Epstein-Barr virus-related immunoproliferative disease No GVHD unresponsive to prior high-dose immunosuppressive therapy No concurrent infections involving the intestinal tract such as: Salmonella Shigella Clostridium difficile (toxin positive) Rotavirus Giardia lamblia Cytomegalovirus by shell vial culture

PATIENT CHARACTERISTICS: Age: 5 to 75 Performance status: Not specified Life expectancy: Not specified Hematopoietic: Platelet count adequate Hepatic: Not specified Renal: Not specified Other: Able to swallow oral capsules No persistent vomiting of all oral intake No multiorgan failure No sepsis syndrome, including positive bacterial or fungal cultures within 72 hours of study

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 7 days since prior anti-thymocyte globulin Chemotherapy: Concurrent cyclosporine, methotrexate, tacrolimus, mycophenolate mofetil, or prednisone allowed if plan in place to taper or discontinue Endocrine therapy: See Disease Characteristics Radiotherapy: Not specified Surgery: Not specified Other: At least 7 days since prior investigational agents At least 7 days since prior immunosuppressive agents At least 24 hours since prior drugs that suppress gastric acid secretion (e.g., H2 receptor antagonists or omeprazole) No concurrent drugs that suppress gastric acid secretion

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-07; Primary Completion 2002-07 (Actual); Study Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hockenbery, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States